CLINICAL TRIAL: NCT00590720
Title: A Phase 2A, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety and Effect on Exercise Challenge Testing of Multiple Fixed Subcutaneous Doses of MEDI-528, A Humanized Anti-Interleukin-9 Monoclonal Antibody, in Adults With Stable Asthma and Exercise-Induced Bronchoconstriction
Brief Title: A Phase 2A Study to Evaluate the Safety and Effect on Exercise Challenge Testing of MEDI-528 in Adults With Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study is replaced by MI-CP198 per CPM.
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP143
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Results first posted 2014-03-21 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-02

CONDITIONS: Asthma
Keywords: Asthma; Bronchitis
MeSH Terms: conditions — Asthma; Bronchitis | interventions — enokizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MEDI528 50 mg (Experimental): MEDI-528 at a dose of 50 mg administered as a subcutaneous injection twice weekly for 4 weeks
  Interventions: Biological: MEDI528 50 mg
- PLACEBO (Placebo Comparator): Placebo administered as a subcutaneous injection twice weekly for 4 weeks
  Interventions: Other: PLACEBO

INTERVENTIONS:
Biological: MEDI528 50 mg — MEDI-528 at a dose of 50 mg administered as a subcutaneous injection twice weekly for 4 weeks
  Arms: MEDI528 50 mg
Other: PLACEBO — Placebo administered as a subcutaneous injection twice weekly for 4 weeks
  Arms: PLACEBO

SUMMARY:
The main objective of this study is to evaluate the safety and tolerability of multiple fixed doses of MEDI-528 in adult patients with stable asthma and exercise-induced bronchoconstriction (EIB).

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of multiple fixed escalating SC doses of MEDI-528 in adult patients with stable asthma and exercise-induced bronchoconstriction (EIB).

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria:

* Male or female adults, age 18 through 50 years at the time of screening;
* Weight 50-100 kg and body mass index ≤ 35;
* Written informed consent obtained from the patient prior to receipt of any study medication or beginning study procedures;
* Documented clinical history of asthma and receiving stable treatment for ≥ 1 month prior to Study Day 0;
* Airway hyperresponsiveness (AHR) on methacholine inhalation challenge testing at screening (or a documented history within the past 6 months), with provoking concentration of methacholine to cause a 20% fall in FEV1(subscript) (PC20) ≤ 8 mg/mL (Crapo, 2000);
* Exercise-induced bronchoconstriction (EIB) with a decrease in FEV1 (subscript) of ≥ 15% from pre-exercise challenge testing level at screening;
* Able to provide spirometry readings that meet American Thoracic Society (ATS) and European Respiratory Society (ERS) standards (Miller, 2005);
* Women of childbearing potential, unless surgically sterile or at least 1 year post-menopausal, must use two effective methods of avoiding pregnancy (including oral, transdermal, or implanted contraceptives, intrauterine device, female condom, spermicide, diaphragm, cervical cap, abstinence, contraceptive foam, or use of a condom by the sexual partner or sterile sexual partner) from screening through Study Day 0, and must agree to continue using such precautions through Study Day 150. Cessation of birth control after this point should be discussed with a responsible physician. Men, unless surgically sterile, must likewise use an effective method of birth control (condom with spermicide) and must agree to continue using such precautions from screening through Study Day 150;
* Able to complete the study period, including follow-up period, of up to approximately 150 days; and
* Willing to forego other forms of experimental treatment and study procedures during the study and for 30 days after the follow-up period is completed.

Exclusion Criteria:

Patients must have none of the following criteria:

* Receipt of MEDI-528 in any previous clinical study;
* History of allergy or reaction to any component of the study drug formulation;
* Lung disease other than asthma (eg, chronic obstructive pulmonary disease, cystic fibrosis);
* Forced expiratory volume in 1 second (FEV1-subscript) < 70% of predicted values at screening;
* Use of systemic immunosuppressive drugs including systemic corticosteroids, ICS with doses > 800 μg/day budesonide (or another ICS of equivalent dose), long-acting β2 agonists, cromolyn sodium, nedocromil sodium, leukotriene receptor antagonists, theophylline, or omalizumab from screening through Study Day 150;
* Current use of any β-adrenergic antagonist (eg, propranolol);
* Any disease or illness, other than asthma, that is likely to require the use of systemic corticosteroids during the study period;
* Acute illnesses or evidence of significant active infection, such as fever ≥ 38.0°C (100.5°F) from screening through Study Day 0;
* Current allergy vaccination therapy (desensitization immunotherapy);
* Receipt of any investigational drug therapy within 30 days or any biologic(s) within 5 half-lives of the agent prior to screening;
* Pregnancy (women of child bearing potential, unless surgically sterile or at least 1 year postmenopausal, must have a negative serum and urine pregnancy test at screening before methacholine inhalation challenge testing and a negative urine pregnancy test prior to study drug administration on Study Day 0);
* Breastfeeding or lactating woman;
* Evidence of infection with hepatitis B or C virus or HIV-1 or HIV-2, or active infection with hepatitis A; must have negative HIV-1, HIV-2, hepatitis A, B, and C tests at screening;
* History of cancer other than basal cell carcinoma of the skin or cervical carcinoma-in-situ treated with apparent success with curative therapy more than 1 year prior to Study Day 0;
* History of primary immunodeficiency
* History of pancreatitis or currently active gastroduodenal ulcer;
* Current use of tobacco products or a history of use of tobacco products of more than one cigarette per month or equivalent within 1 year prior to randomization or history of smoking of ≥ 10 pack-years;
* History of life-long urinary retention;
* History of anaphylaxis (defined as immediate life-threatening event requiring medical invention);
* Elective surgery planned from screening through Study Day 150;
* Clinically significant abnormality, as determined by the investigator, on 12-lead ECG or chest radiograph at screening;
* History of any disease, evidence of any current disease (other than asthma), any finding upon physical examination, or any laboratory abnormality, that, in the opinion of the investigator or medical monitor, may compromise the safety of the patient in the study or confound the analysis of the study; or
* Any employee of the research site who is involved with the conduct of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Parker, M.D., Study Director — MedImmune LLC
Locations (12):
- United States (9):
  - Institute of Healthcare Assessment, Inc, San Diego, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Waterbury Pulmonary Associates, Waterbury, Connecticut
  - Univ. of South Florida, Asthma, Allergy & Immunology Clinical Research Unit, Tampa, Florida
  - Sneeze,Wheeze & Itch Associates, LLC, Normal, Illinois
  - Northeast Medical Research Associates, Inc, No. Dartmouth, Massachusetts
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Creighton University, Omaha, Nebraska
  - Bernstein Clinical Research Center, Cincinnati, Ohio
- Canada (3):
  - Calgary COPD & Asthma Program, Calgary, Alberta
  - UHN- Toronto Western Hospital, Toronto, Ontario
  - Centre de Recherche Appliquee en Allergie de Quebec, Québec, Quebec

REFERENCES:
- [Derived] Parker JM, Oh CK, LaForce C, Miller SD, Pearlman DS, Le C, Robbie GJ, White WI, White B, Molfino NA; MEDI-528 Clinical Trials Group. Safety profile and clinical activity of multiple subcutaneous doses of MEDI-528, a humanized anti-interleukin-9 monoclonal antibody, in two randomized phase 2a studies in subjects with asthma. BMC Pulm Med. 2011 Feb 28;11:14. doi: 10.1186/1471-2466-11-14. PMID 21356110

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 11 subjects participated in this study from 26Feb2008 to 27Dec2008 at 4 sites in the United States of America.
Pre-assignment Details: Treatment assignments were determined using a block randomization procedure with a 2:1 ratio (MEDI-528:placebo) via an interactive voice response system on Day 0 before study drug administration.
Groups:
- MEDI528 50 mg: MEDI528 at a dose of 50 mg administered as a subcutaneous injection twice weekly for 4 weeks
Period: Overall Study
Arm/Group | PLACEBO | MEDI528 50 mg
Started | 4 | 7
Completed | 3 | 6
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PLACEBO | MEDI528 50 mg | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.8 (13.5) | 32.1 (8.2) | 32.0 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: Number of participants experiencing adverse events (includes both adverse events and serious adverse events)
Time Frame: Days 0 - 150
Population: All participants who received at least one dose of investigational product (MEDI-528 or placebo).
Measure: Number; unit: Participants
Arm/Group | PLACEBO | MEDI528 50 mg
Number analyzed (Participants) | 4 | 7
Participants | 4 | 6

2. Primary Outcome: Incidence of Serious Adverse Events
Description: Number of participants experiencing serious adverse events
Time Frame: Days 0 - 150
Population: All participants who received at least one dose of investigational product (MEDI-528 or placebo).
Measure: Number; unit: Participants
Arm/Group | PLACEBO | MEDI528 50 mg
Number analyzed (Participants) | 4 | 7
Participants | 0 | 1

3. Secondary Outcome: Incidence of Anti-drug Antibodies (ADA) to MEDI-528
Description: Number of participants with ADA to MEDI-528
Time Frame: Days 0, 28, 56, 119, and 150
Population: All participants who received at least one dose of MEDI-528.
Measure: Number; unit: Participants
Arm/Group | PLACEBO | MEDI528 50 mg
Number analyzed (Participants) | 0 | 7
Participants |  | 0

4. Secondary Outcome: Absolute Maximum Change in Forced Expiratory Volume in 1 Second (FEV1)
Description: The clinical activity of MEDI-528 on exercise-induced bronchoconstriction was measured by exercise challenge testing expressed as the maximum change in FEV1 measured before and after exercising on Day 28.
Time Frame: Day 28 (15 minutes prior to exercise and 5, 10, 15, 20, and 30 minutes after exercise)
Population: All participants who received at least 4 doses of investigational product (MEDI-528 or placebo; n=10, 3 placebo and 7 MEDI-528) and performed acceptable spirometry (n=9, with 2 placebo and 7 MEDI-528).
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | PLACEBO | MEDI528 50 mg
Number analyzed (Participants) | 2 | 7
Liter | -0.43 (0.23) | -0.21 (0.39)
Statistical Analysis 1: Comparison: PLACEBO vs MEDI528 50 mg; Test type: Superiority or Other; p = 0.40, Two-sample t-test

5. Secondary Outcome: Absolute Maximum Change in Forced Expiratory Volume in 1 Second (FEV1)
Description: The clinical activity of MEDI-528 on exercise-induced bronchoconstriction was measured by exercise challenge testing expressed as the maximum change in FEV1 before and after exercise on Day 56.
Time Frame: Day 56 (15 minutes prior to exercise and 5, 10, 15, 20, and 30 minutes after exercise)
Population: All participants who received at least 4 doses of investigational product (MEDI-528 or placebo; n=10, 3 placebo and 7 MEDI-528) and had available data (n=8, 2 placebo and 6 MEDI-528).
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | PLACEBO | MEDI528 50 mg
Number analyzed (Participants) | 2 | 6
Liter | -0.60 (0.04) | -0.02 (0.06)
Statistical Analysis 1: Comparison: PLACEBO vs MEDI528 50 mg; Test type: Superiority or Other; p < 0.01, Two-sample t-test

6. Secondary Outcome: Absolute Maximum Change in Forced Expiratory Volume in 1 Second (FEV1)
Description: The clinical activity of MEDI-528 on exercise-induced bronchoconstriction was measured by exercise challenge testing expressed as the maximum change in FEV1 before and after exercise on Day 150.
Time Frame: Day 150 (15 minutes prior to exercise and 5, 10, 15, 20, and 30 minutes after exercise)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | PLACEBO | MEDI528 50 mg
Number analyzed (Participants) | 2 | 6
Liter | -0.54 (0.62) | -0.13 (0.11)
Statistical Analysis 1: Comparison: PLACEBO vs MEDI528 50 mg; Test type: Superiority or Other; p = 0.53, Two-sample t-test

7. Secondary Outcome: Percent Maximum Change in Forced Expiratory Volume in 1 Second (FEV1)
Description: The clinical activity of MEDI-528 on exercise-induced bronchoconstriction was measured by exercise challenge testing expressed as the percent maximum change in FEV1 before and after exercise on Day 28.
Time Frame: Day 28 (15 minutes prior to exercise and 5, 10, 15, 20, and 30 minutes after exercise)
Population: All participants who received at least 4 doses of investigational product (MEDI-528 or placebo; n=10, 3 placebo and 7 MEDI-528) and performed acceptable spirometry (n=9, 2 placebo and 7 MEDI-528).
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | PLACEBO | MEDI528 50 mg
Number analyzed (Participants) | 2 | 7
Percent change | -12.6 (1.53) | -6.49 (11.73)
Statistical Analysis 1: Comparison: PLACEBO vs MEDI528 50 mg; Test type: Superiority or Other; p = 0.22, Two-sample t-test

8. Secondary Outcome: Percent Maximum Change in Forced Expiratory Volume in 1 Second (FEV1)
Description: The clinical activity of MEDI-528 on exercise-induced bronchoconstriction was measured by exercise challenge testing expressed as the percent maximum change in FEV1 before and after exercise on Day 56.
Time Frame: Day 56 (15 minutes prior to exercise and 5, 10, 15, 20, and 30 minutes after exercise)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | PLACEBO | MEDI528 50 mg
Number analyzed (Participants) | 2 | 6
Percent change | -20.1 (7.41) | -1.01 (2.22)
Statistical Analysis 1: Comparison: PLACEBO vs MEDI528 50 mg; Test type: Superiority or Other; p = 0.16, Two-sample t-test

9. Secondary Outcome: Percent Maximum Change in Forced Expiratory Volume in 1 Second (FEV1)
Description: The clinical activity of MEDI-528 on exercise-induced bronchoconstriction was measured by exercise challenge testing expressed as the percent maximum change in FEV1 before and after exercise on Day 150.
Time Frame: Day 150 (15 minutes prior to exercise and 5, 10, 15, 20, and 30 minutes after exercise)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | PLACEBO | MEDI528 50 mg
Number analyzed (Participants) | 2 | 6
Percent change | -15.2 (15.48) | -5.04 (3.91)
Statistical Analysis 1: Comparison: PLACEBO vs MEDI528 50 mg; Test type: Superiority or Other; p = 0.52, Two-sample t-test

10. Secondary Outcome: Area Under the Curve (AUC) of Forced Expiratory Volume in 1 Second (FEV1)
Description: AUC of FEV1 at Day 28
Time Frame: Day 28 (15 minutes prior to exercise and 5, 10, 15, 20, and 30 minutes after exercise)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Liter x min
Arm/Group | PLACEBO | MEDI528 50 mg
Number analyzed (Participants) | 2 | 6
Liter x min | 92.69 (41.14) | 86.04 (15.62)

11. Secondary Outcome: Area Under the Curve (AUC) of Forced Expiratory Volume in 1 Second (FEV1)
Description: AUC of FEV1 at Day 56
Time Frame: Day 56 (15 minutes prior to exercise and 5, 10, 15, 20, and 30 minutes after exercise)
Population: All participants who received at least 4 doses of investigational product (MEDI-528 or placebo; n=10, 3 placebo and 7 MEDI-528) and had available data (n=7, 2 placebo and 5 MEDI-528).
Measure: Mean (Standard Deviation); unit: Liter x min
Arm/Group | PLACEBO | MEDI528 50 mg
Number analyzed (Participants) | 2 | 5
Liter x min | 85.38 (44.72) | 83.35 (22.66)

12. Secondary Outcome: Area Under the Curve (AUC) of Forced Expiratory Volume in 1 Second (FEV1)
Description: AUC of FEV1 at Day 150
Time Frame: Day 150 (15 minutes prior to exercise and 5, 10, 15, 20, and 30 minutes after exercise)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Liter x min
Arm/Group | PLACEBO | MEDI528 50 mg
Number analyzed (Participants) | 2 | 5
Liter x min | 82.53 (18.31) | 81.37 (19.93)

13. Secondary Outcome: Time to Return in Minutes to 90 Percent of Baseline Forced Expiratory Volume in 1 Second (FEV1)
Description: Time to return in minutes to 90 percent of baseline FEV1 (prior to exercise) after 30 minues of exercise on Day 28
Time Frame: Day 28 (15 minutes prior to exercise and 5, 10, 15, 20, and 30 minutes after exercise)
Population: All participants who received at least 4 doses of investigational product (MEDI-528 or placebo; n=10, 3 placebo and 7 MEDI-528) and had available data (n=9, 2 placebo and 7 MEDI-528).
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | PLACEBO | MEDI528 50 mg
Number analyzed (Participants) | 2 | 7
Minutes | 10.00 (0.00) | 5.71 (1.89)

14. Secondary Outcome: Time to Return in Minutes to 90 Percent of Baseline Forced Expiratory Volume in 1 Second (FEV1)
Description: Time to return in minutes to 90 percent of baseline FEV1 (prior to exercise) after exercise on Day 56
Time Frame: Day 56 (15 minutes prior to exercise and 5, 10, 15, 20, and 30 minutes after exercise)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | PLACEBO | MEDI528 50 mg
Number analyzed (Participants) | 2 | 6
Minutes | 10.00 (0.00) | 5.00 (0.00)

15. Secondary Outcome: Time to Return in Minutes to 90 Percent of Baseline Forced Expiratory Volume in 1 Second (FEV1)
Description: Time to return in minutes to 90 percent of baseline FEV1 (prior to exercise) after exercise on Day 150
Time Frame: Day 150 (15 minutes prior to exercise and 5, 10, 15, 20, and 30 minutes after exercise)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | PLACEBO | MEDI528 50 mg
Number analyzed (Participants) | 2 | 6
Minutes | 7.50 (3.54) | 5.00 (0.00)

16. Secondary Outcome: Mean Trough Concentration (Cmin)
Description: Cmin of MEDI-528
Time Frame: Days 0, 3, 7, 10, 14, 17, 21, 24, 28, 32, 37, 42, 56, 70, 84, 119, and 150
Population: All participants who received at least one dose of MEDI-528.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | PLACEBO | MEDI528 50 mg
Number analyzed (Participants) | 0 | 7
Microgram per milliliter |  | 2.207 (1.694)

17. Secondary Outcome: Mean Trough Concentration at Last Measurable Time Point (Cmin_last)
Description: Cmin_last of MEDI-528
Time Frame: Days 0, 3, 7, 10, 14, 17, 21, 24, 28, 32, 37, 42, 56, 70, 84, 119, and 150
Population: All participants who received at least one dose of MEDI-528.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | PLACEBO | MEDI528 50 mg
Number analyzed (Participants) | 0 | 7
Microgram per milliliter |  | 18.123 (10.456)

18. Secondary Outcome: Half-life (T1/2)
Description: T1/2 of MEDI-528
Time Frame: Days 0, 3, 7, 10, 14, 17, 21, 24, 28, 32, 37, 42, 56, 70, 84, 119, and 150
Population: All participants who received at least one dose of MEDI-528.
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | PLACEBO | MEDI528 50 mg
Number analyzed (Participants) | 0 | 7
Day |  | 34.708 (7.891)

19. Secondary Outcome: Accumulation Index
Description: Ratio of trough concentrations after first (Day 0) and last (Day 24) dose of MEDI-528
Time Frame: Days 0 and 24
Population: All participants who received at least one dose of MEDI-528 (n=7) and had available data (n=5).
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | PLACEBO | MEDI528 50 mg
Number analyzed (Participants) | 0 | 5
Ratio |  | 7.615 (5.215)

ADVERSE EVENTS:
Arm/Group | PLACEBO | MEDI528 50 mg
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/7
Other Adverse Events (participants affected / at risk) | 4/4 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=4) | MEDI528 50 mg (N=7)
Nuclear magnetic resonance imaging abnormal (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=4) | MEDI528 50 mg (N=7)
Cyst (General disorders) | 0 (0) | 1 (1)
Injection site irritation (General disorders) | 1 (2) | 1 (2)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood bicarbonate increased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 2 (3)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hyposmia (Nervous system disorders) | 1 (1) | 0 (0)
Nerve root compression (Nervous system disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.